CLINICAL TRIAL: NCT03792737
Title: A Prospective, Multi-center, Randomized Controlled Study Evaluating the Efficacy and Safety of Two Types of Absorbable Surgical Sutures in the Suturing of Thyroid Surgery Incision
Brief Title: A Study of Two Types of Absorbable Surgical Sutures in the Suturing of Thyroid Surgery Incision
Acronym: Nautilus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESC-201702
Record Dates: First submitted 2018-11-29; First posted 2019-01-03 (Actual); Results first posted 2021-01-29 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-02

CONDITIONS: Sutures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational group 1 (Experimental): Investigational group 1: Use the study device Spiral PDS Plus for continuous suture of the ribbon muscles, VICRYL Plus for interrupted suture of the platysma, and MONOCRYL Plus for continuous subcuticular suture.
  Interventions: Device: Spiral PDS Plus; Device: MONOCRYL Plus; Device: VICRYL Plus
- Investigational group 2 (Experimental): Investigational group 2: Use PDS Plus for continuous suture of the ribbon muscles, VICRYL Plus for interrupted suture of the platysma, and the study device Spiral MONOCRYL Plus for continuous subcuticular suture.
  Interventions: Device: Spiral MONOCRYL Plus; Device: PDS Plus; Device: VICRYL Plus
- Control group (Active Comparator): Control group: Use the control device PDS Plus for continuous suture of the ribbon muscles, VICRYL Plus for interrupted suture of the platysma, and the control device MONOCRYL Plus continuous subcuticular suture.
  Interventions: Device: PDS Plus; Device: MONOCRYL Plus; Device: VICRYL Plus

INTERVENTIONS:
Device: Spiral PDS Plus — The Spiral PDS Plus is an antibacterial monofilament, synthetic absorbable device. It contains triclosan, a broad spectrum antibacterial agent. The device consists of barbed suture material, armed with a surgical needle on one end and a fixation loop at the opposite end. The device is designed to anchor with a closed loop at one end and a unidirectional barbed section on the other end. Spiral PDS Plus barbs are oriented in one direction to allow tissue approximation without the need to tie surgical knots.
  Arms: Investigational group 1
Device: Spiral MONOCRYL Plus — The Spiral MONOCRYL Plus is an antibacterial monofilament, synthetic absorbable device. It contains triclosan, a broad spectrum antibacterial agent. The device consists of barbed suture material, armed with a surgical needle on one end and a fixation loop at the opposite end. The device is designed to anchor with a closed loop at one end and a unidirectional barbed section on the other end. Spiral MONOCRYL Plus barbs are oriented in one direction to allow tissue approximation without the need to tie surgical knots.
  Arms: Investigational group 2
Device: PDS Plus — PDS Plus is a non-barbed antibacterial monofilament, synthetic absorbable suture. The suture contains triclosan, a broad spectrum antibacterial agent.
  Arms: Control group; Investigational group 2
Device: MONOCRYL Plus — MONOCRYL Plus is a non-barbed antibacterial monofilament, synthetic absorbable suture. The suture contains triclosan, a broad spectrum antibacterial agent.
  Arms: Control group; Investigational group 1
Device: VICRYL Plus — VICRYL Plus antibacterial suture is a non-barbed synthetic absorbable sterile, surgical suture. The suture contains triclosan, a broad spectrum antibacterial agent.

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of two types of absorbable surgical sutures -- STRATAFIX Spiral PDS Knotless Plus Tissue Control Device and STRATAFIX Spiral MONOCRYL Plus Knotless Tissue Control Device (hereinafter referred to as Spiral PDS Plus and Spiral MONOCRYL Plus) used in thyroid surgery to suture surgical incision.

DETAILED DESCRIPTION:
This study adopts a multicenter, prospective, randomized controlled design. The study population are subjects who undergo thyroid surgery.

Before the surgery, subjects are randomized in 1:1:1 ratio to the investigational group 1 (using Spiral PDS Plus), investigational group 2 (using Spiral MONOCRYL Plus) and control group. See the table below for the specific suture levels, materials and techniques of each group.

A blinded central imaging evaluation will be performed on the healing condition of surgical incision on Day 5-7 post-surgery. The subjects will be blinded to the type of suture used for wound closure.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is ≥18, and <70 years old
2. Planned open thyroid surgery, adopting an anterior cervical curved incision (Kocher's incision);
3. Subject who volunteers to participate in this study, follows the study requirements and follow-up visit and signs the written Informed Consent Form voluntarily;
4. Subject who agrees to not schedule any elective surgical operation except the study surgery before the study is completed;
5. The investigator considers the subject's expected postoperative survival time is not less than 3 months.

Exclusion Criteria:

1. Female subjects who are pregnant or lactation at screening;
2. Preoperative clinical staging shows stage IV thyroid cancer, or cervical lymph nodes dissection is planned;
3. Suspected or confirmed anaplastic thyroid cancer;
4. Peripheral vascular disease affecting blood supply of the neck;
5. Active infectious collagenosis (e.g. scleroderma), or any other disease that would interfere with wound healing;
6. Fasting plasma glucose ≥7.7 mmol/L;
7. History of coagulation diseases;
8. Current oral or intravenous antibiotic therapy for existing disease or infection;
9. History of immunosuppressant use (e.g. steroids) within the last 6 months;
10. Chemotherapy or radiotherapy within the last 6 months, or planned chemotherapy or radiotherapy during the study;
11. Personal or family history of keloid formation or hyperplasia;
12. Current participation in any other drug (within 30 days or within 5 half-lives of the investigational drug) or device clinical study;
13. History of any thyroid surgery, except thyroid fine-needle aspiration biopsy;
14. Planned use of skin adhesive at the incision site;
15. The subject is not suitable for participating in this study for any other reasons, as judged by the investigator.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zhang, Principal Investigator — First Hospital of China Medical University
Locations (10):
- China (10):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical college Huazhong University of science and technologyUnion Hospital Tongji Medical college Huazhong University of science and technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'An Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University, Beijing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: one subject didn't participate screen visit and randomize, but receive IP(group 2) treatment by mistake. investigator collect his safety information. so in protocol enrollment plan is 501 subjects, but actually received screen and randomization is 500 patients.
Groups:
- Investigational Group 1: Spiral PDS Plus
- Investigational Group 2: Spiral MONOCRYL Plus
- Control groupEdit: PDS Plus or Monocryl Plus
Period: Overall Study
Arm/Group | Investigational Group 1 | Investigational Group 2 | Control groupEdit
Started (Participated in randomization) | 166 | 167 | 167
Safety Analysis Set (subjects who received investigational product treatment and had post-baseline follow-up data) | 162 | 161 (one subject didn't participate screen visit or randomize, but receive IP treatment by mistake.) | 162
Full Analysis Set (Subjects who were randomized and received corresponding investigational product(IP) treatment, with at least one data to evaluate the post-baseline effectiveness.) | 162 | 160 | 162
Completed (Completed all the study visits) | 160 | 159 | 158
Not Completed | 6 | 8 | 9

BASELINE CHARACTERISTICS:
Population: Full Analysis Population(FAS): FAS consists of all the enrolled subjects who were randomized and at least post-baseline effectiveness endpoint evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Group 1 | Investigational Group 2 | Control groupEdit | Total
Number analyzed (Participants) | 162 | 160 | 162 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.66) | 41.2 (10.84) | 40.3 (11.32) | 40.5 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 118 | 111 | 336
  Male | 55 | 42 | 51 | 148
Race/Ethnicity, Customized [Number; unit: Participants]
  Han | 158 | 157 | 155 | 470
  Other | 4 | 3 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Wound Healing Grade
Description: Percentage of Participants with Grade A Healing of Surgical Incision
Time Frame: 5-7days
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Investigational group1: Spiral PDS Plus
- Investigational group2: Spiral MONOCRYL Plus
- Control Group: PDS Plus or Monocryl Plus
Arm/Group | Investigational group1 | Investigational group2 | Control Group
Number analyzed (Participants) | 154 | 157 | 156
percentage | 99.35 [96.44 to 99.98] | 98.73 [95.47 to 99.85] | 99.36 [96.48 to 99.98]

2. Secondary Outcome: Incision Closure Time
Description: the time required from the first needle insertion for stitching ribbon muscles to the completion of intradermal suture (minutes)
Time Frame: during surgery, an average of around 12 Mins
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Investigational group1 | Investigational group2 | Control Group
Number analyzed (Participants) | 162 | 160 | 162
minutes | 11.285 (3.2635) | 11.198 (3.1298) | 11.634 (3.4327)

3. Secondary Outcome: Postoperative Incisional Pain Score (Visual Analogue Scale, VAS)
Description: For the postoperative incisional pain score, a score of 0 means no pain, and a score of 10 means unbearable: severely affects sleep with other symptoms, or passive position.
Time Frame: 5-7 Days after Surgery and 28-35 Days after Surgery
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Investigational group1 | Investigational group2 | Control Group
Number analyzed (Participants) | 162 | 160 | 162
Units
  VAS Scale-Visit 4 (5-7 Days after Surgery) | 1.5 (1.49) | 1.5 (1.61) | 1.4 (1.39)
  VAS Scale-Visit 5 (28-35 Days after Surgery) | 0.45 (0.775) | 0.63 (0.991) | 0.66 (1.319)

4. Secondary Outcome: Modified Hollander Wound Evaluation Scale - FAS
Description: Total cosmetic score. Assessed by Central Imaging evaluators using incision pictures to evaluate healing status. range is from 0 to 5, 0 is best and 5 is worst
Time Frame: 28-35 days
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Investigational group1 | Investigational group2 | Control Group
Number analyzed (Participants) | 160 | 159 | 162
scores on a scale | 0.2 (0.53) | 0.1 (0.38) | 0.1 (0.45)

5. Secondary Outcome: Health Related Quality of Life Scale (EQ-5D-5L)
Description: Summary of European Quality of Life-5 Dimensions, 5 Levels Scale (EQ-5D-5L) Index Values by Follow-Up Visit - Full Analysis Set. it's to evaluate subjects Health related quality of life. rang is 0 to 1, 0 is better and 1 is worse
Time Frame: 5-7 days after surgery
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Investigational group1 | Investigational group2 | Control Group
Number analyzed (Participants) | 160 | 160 | 160
scores on a scale | 0.8627 (0.11007) | 0.8537 (0.11843) | 0.8489 (0.11648)

6. Secondary Outcome: Health Related Quality of Life Scale (EQ-5D-5L)
Description: Summary of European Quality of Life-5 Dimensions, 5 Levels Scale (EQ-5D-5L) Index Values by Follow-Up Visit - Full Analysis Set. it's to evaluate subjects Health related quality of life. rang is 0 to 1. 0 is better and 1 is worse.
Time Frame: 28-35 days after surgery
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Investigational group1 | Investigational group2 | Control Group
Number analyzed (Participants) | 160 | 159 | 158
scores on a scale | 0.9159 (0.10566) | 0.9024 (0.10738) | 0.9230 (0.10489)

7. Secondary Outcome: Summary of EQ-5D VAS Score
Description: Summary of European Quality of Life-5 Dimensions, 5 Levels Scale (EQ-5D-5L) Index Values by Follow-Up Visit - Full Analysis Set. it's to evaluate subjects Health related quality of life. rang is 0 to 100. 100 is best and 0 is worst.
Time Frame: 5-7 Days after surgery
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Investigational group1 | Investigational group2 | Control Group
Number analyzed (Participants) | 160 | 160 | 160
scores on a scale | 88.1 (10.02) | 87.7 (10.32) | 88.3 (9.45)

8. Secondary Outcome: Summary of EQ-5D VAS Score
Description: Summary of European Quality of Life-5 Dimensions, 5 Levels Scale (EQ-5D-5L) Index Values by Follow-Up Visit - Full Analysis Set. it's to evaluate subjects Health related quality of life. rang is 0 to 100.
Time Frame: 28-35 Days after surgery
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Investigational group1 | Investigational group2 | Control Group
Number analyzed (Participants) | 160 | 159 | 158
scores on a scale | 91.2 (8.95) | 91.7 (7.83) | 92.3 (7.88)

ADVERSE EVENTS:
Time Frame: 35 days
Description: AE is an untoward medical occurrence during the clinical study and which does not necessarily have a causal relationship with the study medical device.
  one subject didn't participate screen visit and randomize, but receive IP(group 2) treatment by mistake. investigator collect his safety information. so the Number of Participants at Risk of group 2 is one more than other rows.
Arm/Group | Investigational Group 1 | Investigational Group 2 | Control groupEdit
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/161 | 0/162
Serious Adverse Events (participants affected / at risk) | 4/162 | 4/161 | 2/162
Other Adverse Events (participants affected / at risk) | 44/162 | 46/161 | 50/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Group 1 (N=162) | Investigational Group 2 (N=161) | Control groupEdit (N=162)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Breast adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — General disorders and administration site conditions
Skin oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Group 1 (N=162) | Investigational Group 2 (N=161) | Control groupEdit (N=162)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 30 (30) | 32 (32) | 31 (31)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (6) | 16 (16) | 16 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 25 (26) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the principal investigator(PI) is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03792737/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT03792737/SAP_000.pdf